CLINICAL TRIAL: NCT00958893
Title: An Open-Label Extension Study Evaluating Safety and Efficacy of Proellex® In Women With Leiomyomata Who Have Previously Completed ZPU 003 Ext
Brief Title: An Extension Study Evaluating Safety and Efficacy of Proellex® In Women Who Have Previously Completed ZPU 003 Ext
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Repros stopped the study for safety and FDA put the study on hold for safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZPU-003 Extension 2
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 25 mg Proellex (Experimental): 25 mg Proellex daily
  Interventions: Drug: 25 mg Proellex

INTERVENTIONS:
Drug: 25 mg Proellex — one 25 mg capsules
  Other Names: CDB-4124; Proellex

SUMMARY:
An open label, extension study for subjects completing the ZPU-003 Ext 1 study.

DETAILED DESCRIPTION:
This is an open label, extension study for subjects completing the ZPU-003 Ext 1 study and an off-drug interval (menses), prior to the start of the first 16-week dosing cycle. Subjects will receive a 50 mg Proellex® daily dose. Total study participation for ZPU-003 Ext 2 (Extension 2) may be up to three 4 month drug cycles separated by off drug intervals.

ELIGIBILITY:
Inclusion Criteria:

* Four subjects at one site whom have completed ZPU 003 Ext 1 study

Exclusion Criteria:

* All other subjects

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (1):
- Advances in Health, Inc., Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 25 mg Proellex
Started | 4
Completed | 0
Not Completed | 4
Not completed — Study prematurely terminated | 4

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated
Arm/Group | 25 mg Proellex
Number analyzed (Participants) | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Further Evaluate Adverse Events of a 25 mg Dose of Proellex® Administered to Women Once Daily for Three 4 Month Cycles Separated by Off-drug Intervals.
Time Frame: three 4 month cycles separated by off-drug intervals
Arm/Group | 25 mg Proellex
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No adverse event data is available.
Arm/Group | 25 mg Proellex
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights